CLINICAL TRIAL: NCT03026764
Title: Patient Satisfaction and Costs Associated With Total Hip Arthroplasty
Brief Title: Inpatient vs Outpatient Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 106362
Record Dates: First submitted 2016-03-09; First posted 2017-01-20 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis
Keywords: cost; total hip replacement; outpatient Surgery; satisfaction; arthroplasty
MeSH Terms: conditions — Osteoarthritis; Personal Satisfaction | interventions — Inosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient (Experimental): Patients in the outpatient group (same day discharge following THA) are discharged the same day following surgery. All patients are required to meet the discharge criteria to be sent home (i.e., capable of using crutches, relatively free of pain, free of nausea and vomiting, free of excess bleeding, alert and oriented, given take-home medications, and in the company of a caregiver).
  Interventions: Procedure: Outpatient
- Inpatient (Active Comparator): Patients in the inpatient group (following day discharge following THA) stay in the hospital overnight and then are discharged home the next day. All patients are required to meet the discharge criteria to be sent home (i.e., capable of using crutches, relatively free of pain, free of nausea and vomiting, free of excess bleeding, alert and oriented, given take-home medications, and in the company of a caregiver).
  Interventions: Procedure: Inpatient

INTERVENTIONS:
Procedure: Outpatient — Patients in the outpatient group will be discharged from the hospital the same day of surgery following a total hip arthroplasty
  Arms: Outpatient
Procedure: Inpatient — Patients in the inpatient group will be discharged from the hospital the following day after a total hip arthroplasty
  Arms: Inpatient

SUMMARY:
This study is a pragmatic randomized clinical trial comparing standard inpatient total hip arthroplasty with same day discharge. Patients who are medically well and have a good support structure at home will be randomized to inpatient or same day discharge. The investigators will compare patient costs from the perspective of the Ministry of Health, the institution, society and the patient. The investigators will also record complications, patient satisfaction, functional ability and quality of life.

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) is currently one of the most successful procedures in orthopaedics. Over the last 40 years, postoperative care has significantly evolved. Initially, the standard procedure following THA was that patients were required to stay in the hospital to recover for 2.5 to 3 weeks. However, with the implementation of less invasive techniques, coupled with early weight bearing and more comprehensive postoperative rehabilitation protocols, inpatient stays have drastically decreased on average to 2 to 3 days. A new, minimally invasive surgical (MIS) technique has led to an even larger decrease in hospital stays, culminating in a same day discharge. The possibility of early mobilization, combined with an increasing push from patients to accelerate recovery and return to activities, have led to the implementation of outpatient THA in select patients. For same day discharge to succeed, extensive preoperative and perioperative care must accompany the procedure. Furthermore, more aggressive rehabilitation and improved pain control is crucial for successful outpatient THA. For younger patients that need to return to work as early as possible, a quicker recovery time is essential. Perfecting outpatient THA is a crucial step towards achieving these requirements.

There are 4 major components to a successful THA: pain relief, functional recovery, patient satisfaction and durable reconstruction. Outpatient THA is a fairly new concept in arthroplasty, and patient satisfaction has not been properly assessed following this new THA protocol. Satisfaction in accordance with THA refers to a patient achieving their functional and pain expectations. A similar study evaluating patient satisfaction of a randomized control trial (RCT) of inpatient versus outpatient anterior cruciate ligament (ACL) reconstructions reported that outpatient satisfaction following surgery is higher than inpatient satisfaction. Although this is a different procedure, it would seem outpatient ACL reconstruction and outpatient THA has similar pain levels, safety and patient satisfaction. The goal with outpatient surgery with regards to satisfaction is providing patients with relief of their anxiety, while allowing them earlier control of their independence. Potential advantages of outpatient surgery include that patients are permitted to recover in a secure, private and comfortable home environment, while surgeons will improve efficiency and time management with the decreased responsibilities of having to visit their inpatients.

In addition to the potential satisfaction benefit, outpatient THA is a potential source of cost savings for both the patient and the hospital. Numerous efforts by hospitals have been made to decrease costs and increase available beds for additional patients. A previous study investigating the financial effects of outpatient THA found that the average hospital bill for outpatients was $4000 less than for the inpatients. Including preoperative physical therapy and home healthcare, the total charges for outpatients was $2500 less than inpatients. A similar study demonstrated that select individuals can successfully undergo THA in an outpatient setting with no increase in complications, while also receiving a substantial savings to the patient and the healthcare system. By reducing costs and increasing healthcare staff availability, hospitals can allocate more money to areas in need of funding, while wait times can drastically reduce for future patients.

The most important part of preoperative care for a successful outpatient THA is giving the patient appropriate goals and expectations. Patients should be educated by the anaesthesiology team, the physical and occupational therapist, the surgeon, the nurses, and anyone else involved in the surgery. Patients are required to attend classes explaining the various aspects of the operative experience, as well as discharge goals and techniques for postoperative home rehabilitation. Furthermore, functional and symptomatic goals need to be clearly defined. In these educational sessions, pain management strategies are one of the main focuses. To have a successful same day discharge, patients must be well versed in pain management and proper rehabilitation strategies. Before the preoperative class, all patients are instructed to practice certain skills, such as bed transfer, cane/crutches use and gait training. Potential complications are discussed so that the patient is reassured with what is normally supposed to happen following surgery. The goal of preoperative care is that the patient has a defined set of goals and expectations for their surgery, medications, and rehabilitation.

For outpatient THA surgery, it is preferred to perform the surgery in the morning to facilitate same day discharge. Immediately following surgery, the primary goals are to treat pain, nausea and hypovolemia. Prior to symptoms arriving, these issues have to be dealt with using the proper fluids and medications. Physical therapy is usually initiated 3 to 4 hours following surgery. The combination of this early rehabilitation program, combined with the minimally invasive surgical technique is vital to the rapid recovery process. Home physical therapy should begin immediately, with a focus on ambulation. The patient is then asked for a follow-up visit within 1 week of the surgery to make sure all of the patient's goals have been met.

The primary concern with outpatient THA is safety of the patient. There are also concerns including emergency room readmissions in patients who have difficulty once home in the immediate postoperative period. Furthermore, some patients will require transfer to an inpatient facility when they are experiencing a delayed recovery after surgery.

Anecdotal data was collected prior to the start of this research project. Since there was a clinical practice change, informal conversations with outpatient THA demonstrated that 10/11 patients would have outpatient surgery again, and 9/11 would recommend outpatient THA surgery to others. These encouraging findings are an important justification for performing the present study.

Although previous THA outpatient studies have demonstrated successful results, it is imperative to complete a RCT to diminish any bias associated with these findings. In the absence of high quality comparative evidence, the success in same day discharge THA may be a result of selection bias, since previous research is largely driven by observational studies of highly selected populations. This would severely decrease the generalizability of previous studies. To our knowledge, this will be the first level one study that will investigate the cost, early complications and patient satisfaction associated with outpatient THA in a pragmatic selection of patients. This study will answer important questions on how to best treat patients undergoing THA, and whether an earlier discharge following surgery affects patient outcomes.

A retrospective analysis of over 50,000 THA and TKA procedures found no differences in 30-day major complications or readmissions among patients with a zero to two-day hospital stay compared to those discharged on day three or four postoperative. The rate of serious adverse events in the inpatient group is expected to be greater than five percent. To define a non-inferiority margin we agreed that no more than a five percent increase in the risk of serious adverse event (RD ≥ 6% favoring inpatient care) was acceptable. If the risk in the inpatient group ranges between five to eight percent and there is truly no difference in risk of serious adverse event between the groups, then a maximum of 506 patients are required to be 80% certain that the upper limit of a one-sided 95% confidence interval will exclude a difference in favour of the inpatient group of more than six percent. Given that the primary outcome is being measured at 3-months postoperative, we anticipate a low lost-to-follow-up rate. Previous studies conducted at the study site in similar patients demonstrate loss to follow up rates less than one percent for the first 3 months. Therefore, to account for a potential one percent dropout rate we inflated our sample size to 511.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiologists (ASA) score equal to or less than 3
2. Have the ability to read and understand English (printed instructions are provided in English only)
3. Live within a 60 minute driving distance of University Hospital (UH)
4. Home / cell phone access
5. An adult to accompany patient home post-operatively
6. Sufficient caregiver support

Exclusion Criteria:

1. Patient has significant pain management issues
2. Patient / family history of anesthesia related complication(s) (e.g., malignant hyperthermia, pseudocholinesterase deficiency, airway difficulties, obstructive sleep apnea)
3. Obesity that significantly impacts the patient's ability to mobilize
4. Anaphylaxis to penicillin
5. Significant psycho / social issues that would prevent the patient from managing at home safely
6. Cognitive issues that preclude the ability to understand instructions
7. Lack of an appropriate social network that can observe the patient post-operatively

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Indirect and Direct Costs of Treatment | 3 months
  ER visits, clinician visits, caregiver lost productivity, tests, etc
Early complications and adverse events | 3 months
  falls, wound problems, pulmonary embolism, deep vein thrombosis, infection, etc
Standardized measure of health outcome (EQ-5D) | 3 months
  utility

SECONDARY OUTCOMES:
Patient Satisfaction Questionnaire | 3 months
  Patient satisfaction with care pre, peri and postoperative
Western Ontario McMaster Osteoarthritis Index (WOMAC) | 3 months
  Functional outcome
Harris Hip Score | 3 months
  Functional Outcome
Short Form - 12 | 3 months
  Quality of Life
Pain Numeric Scale Rating | 3 months
  Pain
Caregiver Assistance Scale | 2 weeks
  Caregiver Confidence
Caregiver Strain Index | 2 weeks
  Caregiver Strain

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD, FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aynardi M, Post Z, Ong A, Orozco F, Sukin DC. Outpatient surgery as a means of cost reduction in total hip arthroplasty: a case-control study. HSS J. 2014 Oct;10(3):252-5. doi: 10.1007/s11420-014-9401-0. Epub 2014 Jul 12. PMID 25264442
- [Background] Berger RA. Total hip arthroplasty using the minimally invasive two-incision approach. Clin Orthop Relat Res. 2003 Dec;(417):232-41. doi: 10.1097/01.blo.0000096828.67494.95. PMID 14646722
- [Background] Berger RA, Jacobs JJ, Meneghini RM, Della Valle C, Paprosky W, Rosenberg AG. Rapid rehabilitation and recovery with minimally invasive total hip arthroplasty. Clin Orthop Relat Res. 2004 Dec;(429):239-47. doi: 10.1097/01.blo.0000150127.80647.80. PMID 15577494
- [Background] Berger RA. A comprehensive approach to outpatient total hip arthroplasty. Am J Orthop (Belle Mead NJ). 2007 Sep;36(9 Suppl):4-5. PMID 17948159
- [Background] Bertin KC. Minimally invasive outpatient total hip arthroplasty: a financial analysis. Clin Orthop Relat Res. 2005 Jun;(435):154-63. doi: 10.1097/01.blo.0000157173.22995.cf. PMID 15930933
- [Background] Charnley J. Present status of total hip replacement. Ann Rheum Dis. 1971 Nov;30(6):560-4. doi: 10.1136/ard.30.6.560. No abstract available. PMID 5130137
- [Background] Dorr LD, Maheshwari AV, Long WT, Wan Z, Sirianni LE. Early pain relief and function after posterior minimally invasive and conventional total hip arthroplasty. A prospective, randomized, blinded study. J Bone Joint Surg Am. 2007 Jun;89(6):1153-60. doi: 10.2106/JBJS.F.00940. PMID 17545416
- [Background] Dorr LD, Thomas D, Long WT, Polatin PB, Sirianni LE. Psychologic reasons for patients preferring minimally invasive total hip arthroplasty. Clin Orthop Relat Res. 2007 May;458:94-100. doi: 10.1097/BLO.0b013e31803212dc. PMID 17224839
- [Background] Dorr LD, Thomas DJ, Zhu J, Dastane M, Chao L, Long WT. Outpatient total hip arthroplasty. J Arthroplasty. 2010 Jun;25(4):501-6. doi: 10.1016/j.arth.2009.06.005. Epub 2009 Jul 28. PMID 19640672
- [Background] Husted H, Holm G, Jacobsen S. Predictors of length of stay and patient satisfaction after hip and knee replacement surgery: fast-track experience in 712 patients. Acta Orthop. 2008 Apr;79(2):168-73. doi: 10.1080/17453670710014941. PMID 18484241
- [Background] Krywulak SA, Mohtadi NG, Russell ML, Sasyniuk TM. Patient satisfaction with inpatient versus outpatient reconstruction of the anterior cruciate ligament: a randomized clinical trial. Can J Surg. 2005 Jun;48(3):201-6. PMID 16013623
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Background] Lovell TP. Single-incision direct anterior approach for total hip arthroplasty using a standard operating table. J Arthroplasty. 2008 Oct;23(7 Suppl):64-8. doi: 10.1016/j.arth.2008.06.027. PMID 18922376
- [Background] Mears DC, Mears SC, Chelly JE, Dai F, Vulakovich KL. THA with a minimally invasive technique, multi-modal anesthesia, and home rehabilitation: factors associated with early discharge? Clin Orthop Relat Res. 2009 Jun;467(6):1412-7. doi: 10.1007/s11999-009-0785-y. Epub 2009 Mar 20. PMID 19301081
- [Background] Chen D, Berger RA. Outpatient minimally invasive total hip arthroplasty via a modified Watson-Jones approach: technique and results. Instr Course Lect. 2013;62:229-36. PMID 23395028
- [Derived] Zomar BO, Marsh JD, Bryant DM, Lanting BA. The cost of outpatient versus inpatient total hip arthroplasty: a randomized trial. Can J Surg. 2022 Sep 1;65(5):E553-E561. doi: 10.1503/cjs.003821. Print 2022 Sep-Oct. PMID 36302128
- [Derived] Zomar BO, Marsh JD, Lanting BA, Bryant DM. A protocol for a randomized controlled trial investigating the safety and cost-effectiveness of outpatient total hip arthroplasty. BMC Musculoskelet Disord. 2020 Oct 8;21(1):663. doi: 10.1186/s12891-020-03699-z. PMID 33032566